CLINICAL TRIAL: NCT02568111
Title: Brimonidine Tartrate for the Treatment of Injection Related Erythema Associated With Sub-cutaneous Administration of Peginterferon Beta-1a (BRITE)
Brief Title: Brimonidine Tartrate for the Treatment of Injection Related Erythema
Acronym: BRITE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NLD-PEG-14-10784; 2015-002159-89 (EudraCT Number)
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS)
Keywords: erythema; PLEGRIDY; injection site reaction (ISR); MS; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Erythema; Injection Site Reaction | interventions — peginterferon beta-1a; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- brimonidine tartrate (Experimental): Participants will apply gel to injection site erythema area after IRE development post peginterferon beta-1a injection
  Interventions: Drug: peginterferon beta-1a; Drug: brimonidine tartrate
- Vehicle Gel (Placebo Comparator): Participants will apply vehicle gel placebo to injection site erythema area after IRE development post peginterferon beta-1a injection
  Interventions: Drug: peginterferon beta-1a; Drug: Vehicle Gel

INTERVENTIONS:
Drug: peginterferon beta-1a — SC administration as prescribed by the physician- initial dose of 63 μg followed by 94 μg dose on day 15 and 125 μg on day 29
  Other Names: PEGylated Interferon Beta-1a; PEG IFN β-1a; Plegridy; BIIB017
Drug: brimonidine tartrate — Applied to injection site as specified in the treatment arm. Commercially available Mirvaso (Brimonidine tartrate) gel will be provided by Galderma.
  Other Names: Mirvaso
  Arms: brimonidine tartrate
Drug: Vehicle Gel — Matched placebo applied to injection site as specified in the treatment arm. Matching vehicle gel will be provided by Galderma.
  Arms: Vehicle Gel

SUMMARY:
The primary objective of this study is to evaluate the Injection Related Erythema (IRE) mitigation effect of a single administration of brimonidine tartrate in comparison with a vehicle gel (placebo).

The secondary study objectives are to evaluate the IRE mitigation effect of a single administration of brimonidine tartrate in comparison with a vehicle gel on a more stringent definition scale, in accordance with the primary endpoint of the original brimonidine pivotal trials and participants' satisfaction with the overall appearance of their skin.

DETAILED DESCRIPTION:
Participants naïve to treatment with subcutaneous (SC) interferons or oral Disease Modifying Therapy (DMT) who are about to start PLEGRIDY PEN therapy will be screened for participation in this Phase IV trial. Participants will remain on Plegridy therapy as prescribed by their physician. Plegridy will not be provided to participants by Biogen as a part of this study.

ELIGIBILITY:
Key Inclusion Criteria:

* RRMS patients naïve to treatment with SC interferon or oral and/or IV DMT for which PLEGRIDY is deemed necessary by the treating physician.
* Patient willing and able to complete PSA and PAA questionnaires with minimal assistance.

Key Exclusion Criteria:

* Known allergy to any interferon or any component of peginterferon beta-1a.
* Patients with hypersensitivity to Brimonidine topical gel.
* Patients with other skin disorders.
* History of previous treatment with Brimonidine tartrate.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in either Clinician's Erythema Assessment (CEA) or Patient Erythema Self-Assessment (PSA) scale measured as at least 1-grade improvement on CEA and/or at least 1-grade improvement on PSA scale assessed by the physician and participant | Before and after 6 hours of gel application
  Investigator will evaluate participant's erythema (redness) at the site of injection on a scale of 0 (clear) to 4 (severe) with higher scores indicating higher levels of erythema. Participants rate erythema at the site of injection on a scale of 0 (clear) to 4 (severe) with higher scores indicating higher levels of erythema.

SECONDARY OUTCOMES:
Composite change in both CEA and PSA scale measured as at least 1-grade improvement on CEA and 1-grade improvement on PSA respectively | Before and after 6 hours of gel application
  This composite endpoint is considered to be sensitive enough and directly correlated with participants' satisfaction therapy outcomes.
Composite change in both CEA and PSA scale measured as at least 2-grade improvement on CEA and 2-grade improvement on PSA | Before and after 6 hours of gel application
Participant's self-assessment of satisfaction with the overall appearance of their skin by using a Patient's Assessment of Appearance (PAA) grading scale | Before and after 6 hours of gel application
  PAA satisfaction score will describe how satisfied the participants are with the overall appearance of skin on a scale of 0 (very satisfied) to 4 (very dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen